CLINICAL TRIAL: NCT03431961
Title: Nasal Allergen Challenge - Reproducibility of Biomarkers and Effect of Topical Steroid Treatment
Acronym: NACHO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gail Gauvreau (Other)
Responsible Party: Sponsor-Investigator, Gail Gauvreau, Professor, Hamilton Health Sciences Corporation
Organization: Hamilton Health Sciences Corporation (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: DC002544/HIREB3820
Record Dates: First submitted 2018-02-07; First posted 2018-02-13 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Allergic Asthma
MeSH Terms: interventions — Triamcinolone Acetonide; Triamcinolone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 0.9% normal saline administered twice daily for 14 days
  Interventions: Drug: Placebo
- Intranasal Corticosteroid (Experimental): Triamcinolone acetonide aqueous nasal spray at a dose of 220 mcg administered twice daily (for a total daily dose of 440 mcg) for 14 days
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide — 220 mcg administered twice daily for 14 days
  Other Names: Nasacort
  Arms: Intranasal Corticosteroid
Drug: Placebo — twice daily for 14 days
  Other Names: 0.9% Normal Saline
  Arms: Placebo

SUMMARY:
Subjects with allergic asthma developing the required nasal symptoms in response to nasal allergen titration during a screening period will be randomized 1:1 to one of 2 cohorts. All subjects will have repeated nasal challenges with allergen. One cohort will have nasal saline challenge as control. One cohort will have intranasal corticosteroid intervention.

DETAILED DESCRIPTION:
Eligible subjects will be randomized 1:1 to Cohort A or Cohort B. Each cohort will undergo 3 nasal challenges, each separated by 3 weeks. Cohort A will undergo 2 nasal allergen challenges, and 1 nasal diluent challenge. TNSS, PNIF, spirometry, and samples of blood, urine and nasal secretions will be collected until 24h post-challenge to assess reproducibility. Cohort B will undergo 3 nasal allergen challenges; one of the challenge will be conducted after 14 days treatment with placebo, and one challenge will be conducted after 14 days treatment with triamcinolone acetonide aqueous nasal spray at a dose of 220 mcg administered twice daily for a total daily dose of 440 mcg. TNSS, PNIF, spirometry, and samples of blood, urine, nasal secretions will be collected until 24h post-challenge to determine reproducibility, and nasal tissue will be collected 24h post-challenge to determine effect of steroid treatment.

ELIGIBILITY:
Inclusion Criteria:

* allergic rhinitis + mild asthma

Exclusion Criteria:

* other respiratory disease
* any medication for treatment of asthma/allergic rhinitis with the exception of infrequent beta-2 agonist.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Cellular inflammation | 24 hours after nasal allergen challenge
  Nasal eosinophils

CONTACTS AND LOCATIONS:
Overall Officials: Gail M Gauvreau, PhD, Principal Investigator — McMaster University
Locations (1):
- Cardio- Respiratory Research Laboratory, Hamilton Health Sciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bauer RN, Xie Y, Beaudin S, Wiltshire L, Wattie J, Munoz C, Alsaji N, Oliveria JP, Ju X, MacLean J, Sommer DD, Keith PK, Satia I, Cusack RP, O'Byrne PM, Sperinde G, Hokom M, Li O, Banerjee P, Chen C, Staton T, Sehmi R, Gauvreau GM. Evaluation of the reproducibility of responses to nasal allergen challenge and effects of inhaled nasal corticosteroids. Clin Exp Allergy. 2023 Nov;53(11):1187-1197. doi: 10.1111/cea.14406. Epub 2023 Oct 4. PMID 37794659